CLINICAL TRIAL: NCT00000225
Title: Alternate-Day Buprenorphine Administration. Phase VI
Brief Title: Alternate-Day Buprenorphine Administration. Phase VI - 7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06969-7; R01-06969-7
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-06

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to determine if four times a subject's daily maintenance dose will hold for 96 hours without changes in agonist and antagonist effects.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1992-12

PRIMARY OUTCOMES:
Drug use
Opioid withdrawal
Opioid agonist effects
Dose identification
Pupil diameter

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] patry, Bickel, Tzanis, Badger (in preparation). Every fourth day dosing with buprenorphine (1) A comparison of four schedules under blind-dosing procedures.. Patry, Bickel, Tzanis, Badger (in preparation). Every fourth day dosing with buprenorphine (1) A comparison of four different dosing schedules under blind-dosing procedures.